CLINICAL TRIAL: NCT01856218
Title: An Open-Label Phase 1/2 Study to Assess the Safety, Efficacy and Dose of UX003 rhGUS Enzyme Replacement Therapy in Patients With Mucopolysaccharidosis Type 7 (MPS 7)
Brief Title: An Open-Label Phase 1/2 Study to Assess the Safety, Efficacy and Dose of Study Drug UX003 Recombinant Human Beta-glucuronidase (rhGUS) Enzyme Replacement Therapy in Patients With Mucopolysaccharidosis Type 7 (MPS 7)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UX003-CL201
Expanded Access: NCT03775174 (Available)
Record Dates: First submitted 2013-05-08; First posted 2013-05-17 (Estimated); Results first posted 2018-01-05 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Mucopolysaccharidosis Type 7
Keywords: Mucopolysaccharidosis type 7, MPS 7, Sly syndrome, enzyme replacement therapy, rare disease, lysosomal storage disease, metabolic disorder
MeSH Terms: conditions — Mucopolysaccharidosis VII; Rare Diseases; Lysosomal Storage Diseases; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (1):
- UX003 (Experimental): During the initial 14-week treatment period of the study, participants receive 2 mg/kg UX003 every other week (QOW) for 12 weeks. At Week 14, participants continue on UX003 therapy and begin a forced dose titration period for an additional 24 weeks at the dose sequence of 1, 4, and 2 mg/kg UX003 QOW as follows: 1 mg/kg UX003 for 8 weeks beginning on Week 14; then 4 mg/kg UX003 for 8 weeks beginning on Week 22; then 2 mg/kg UX003 for 8 weeks beginning on Week 30. Following the 24 week forced dose titration period, participants who continue on treatment (continuation period) received 2 mg/kg UX003 QOW beginning at Week 38 for up to an additional 36 weeks.
  After the first phase of the study, participants who elect to continue drug treatment are transitioned to the long-term extension phase, where they are treated with UX003 at 4 mg/kg beginning at Week 74, for up to an additional 168 weeks.
  Interventions: Drug: UX003

INTERVENTIONS:
Drug: UX003

SUMMARY:
UX003-CL201 is an open-label Phase 1/2 study to assess the safety, efficacy, and dose of UX003 in MPS 7 patients via intravenous (IV) administration every other week (QOW) for 36 weeks with up to an additional 36 weeks from the optional continuation period. Up to 5 participants, who are between 5 and 30 years of age inclusive, will be enrolled and treated with UX003.

The initial 12-week treatment period will be followed by a 24-week forced dose titration period to assess the optimal dose. Participants who complete both the initial treatment and forced dose titration periods will continue treatment in a 36- week continuation period.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of MPS 7 based on leukocyte or fibroblast glucuronidase enzyme assay or genetic testing confirming diagnosis.
* Elevated urinary glycosaminoglycan (uGAG) excretion at a minimum of 2-fold over normal.
* Between 5 and 30 years of age, inclusive (approximately 2 subjects between the ages of 20-30 years).
* Willing and able to provide written, signed informed consent, or in the case of subjects under the age of 18 (or 16 years, depending on the region), provide written assent (if required) and written informed consent by a legally authorized representative after the nature of the study has been explained, and prior to any research-related procedures.
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study.
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study. Females considered not of childbearing potential include those who have had tubal ligation at least one year prior to Screening, or who have had total hysterectomy.

Exclusion Criteria:

* Has undergone a successful bone marrow or stem cell transplant or has any degree of detectable chimaerism with donor cells.
* Any known hypersensitivity to rhGUS or its excipients that, in the judgment of the Investigator, places the subject at increased risk for adverse effects.
* Pregnant or breastfeeding at Screening or planning to become pregnant (self or partner) at any time during the study.
* Use of any investigational product (drug or device or combination) within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments at any time during the study.
* Has a condition of such severity and acuity, in the opinion of the Investigator, that it warrants immediate surgical intervention or other treatment or may not allow safe study participation.
* Has a concurrent disease or condition that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study, or would interfere with study participation or affect safety.

Ages: 5 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2013-11; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Jones, MD, Principal Investigator — Univeristy of Manchester
Locations (1):
- Manchester Academic Health Science Centre, Manchester, United Kingdom

REFERENCES:
- [Derived] Qi Y, McKeever K, Taylor J, Haller C, Song W, Jones SA, Shi J. Pharmacokinetic and Pharmacodynamic Modeling to Optimize the Dose of Vestronidase Alfa, an Enzyme Replacement Therapy for Treatment of Patients with Mucopolysaccharidosis Type VII: Results from Three Trials. Clin Pharmacokinet. 2019 May;58(5):673-683. doi: 10.1007/s40262-018-0721-y. PMID 30467742

RESULTS

PARTICIPANT FLOW:
Groups:
- UX003: During the initial 14-week treatment period of the study, participants received 2 mg/kg UX003 every other week (QOW) for 12 weeks. At Week 14, participants continued on UX003 therapy and began a forced dose titration period for an additional 24 weeks at the dose sequence of 1, 4, and 2 mg/kg UX003 QOW as follows: 1 mg/kg UX003 for 8 weeks beginning on Week 14; then 4 mg/kg UX003 for 8 weeks beginning on Week 22; then 2 mg/kg UX003 for 8 weeks beginning on Week 30. Following the 24 week forced dose titration period, participants who continued on treatment (continuation period) received 2 mg/kg UX003 QOW beginning at Week 38 for up to an additional 36 weeks.
  After the first phase of the study, participants who elected to continue drug treatment were transitioned to the long-term extension phase, where they were treated with UX003 at 4 mg/kg beginning at Week 74, for up to an additional 168 weeks.
Period: First Phase
Arm/Group | UX003
Started | 3
Completed | 3
Not Completed | 0
Period: Long-Term Extension Phase
Arm/Group | UX003
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- UX003: During the initial 14-week treatment period of the study, participants received 2 mg/kg UX003 QOW for 12 weeks. At Week 14, participants continued on UX003 therapy and began a forced dose titration period for an additional 24 weeks at the dose sequence of 1, 4, and 2 mg/kg UX003 QOW as follows: 1 mg/kg UX003 for 8 weeks beginning on Week 14; then 4 mg/kg UX003 for 8 weeks beginning on Week 22; then 2 mg/kg UX003 for 8 weeks beginning on Week 30. Following the 24 week forced dose titration period, participants who continued on treatment (continuation period) received 2 mg/kg UX003 QOW beginning at Week 38 for up to an additional 36 weeks.
  After the first phase of the study, participants who elected to continue drug treatment were transitioned to the long-term extension phase, where they were treated with UX003 at 4 mg/kg beginning at Week 74, for up to an additional 168 weeks.
Arm/Group | UX003
Number analyzed (Participants) | 3
Age, Customized [Count of Participants; unit: Participants]
  Children (2-11 years) | 2
  Adults (18-64 years) | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Urinary Glycosaminoglycan (uGAG) Dermatan Sulfate
Description: Percentage change from baseline in the concentration of uGAGs normalized to the urinary creatinine concentration as measured by liquid chromatography-mass spectrometry/mass spectrometry-dermatan sulfate.
Time Frame: Baseline, Week 14, Week 22, Week 30, Week 38, Week 72, and end of study (up to Week 132)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | UX003
Number analyzed (Participants) | 3
percentage change
  Initial treatment-Week 14 | -50.41 (7.895)
  Forced dose titration-Week 22 | -38.94 (7.137)
  Forced dose titration-Week 30 | -63.49 (6.889)
  Forced dose titration-Week 38 | -51.82 (9.033)
  Continuation-Week 72 | -54.2 (8.442)
  Long term extension-end of study | -34.44 (48.56)

2. Primary Outcome: Percentage Change From Baseline in uGAG Chondroitin Sulfate
Description: Percentage change from baseline in the concentration of uGAGs normalized to the urinary creatinine concentration as measured by liquid chromatography-mass spectrometry/mass spectrometry-chondroitin sulfate.
Time Frame: Baseline, Week 14, Week 22, Week 30, Week 38, Week 72, and end of study (up to Week 132)
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | UX003
Number analyzed (Participants) | 3
percentage change
  Initial treatment-Week 14 | -52.5 (13.726)
  Forced dose titration-Week 22 | -47.58 (3.958)
  Forced dose titration-Week 30 | -60.78 (7.207)
  Forced dose titration-Week 38 | -52.08 (13.298)
  Continuation-Week 72 | -56.96 (13.379)
  Long term extension-end of study | -30.83 (40.794)

3. Primary Outcome: Number of Participants With Any ≥ 50% Decrease in uGAG
Description: Participants with a ≥ 50% decrease in the concentration of uGAGs normalized to the urinary creatinine concentration as measured by liquid chromatography-mass spectrometry/mass spectrometry-dermatan sulfate or chondroitin sulfate.
Time Frame: up to Week 132
Measure: Count of Participants; unit: Participants
Arm/Group | UX003
Number analyzed (Participants) | 3
Participants | 3

4. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), Deaths, and Study/Treatment Discontinuations
Description: Adverse Event (AE): any untoward medical occurrence in a subject, whether or not considered drug related. SAE: an AE or suspected adverse reaction that at any dose results in any of the following outcomes: death; a life-threatening AE; inpatient hospitalization or prolongation of existing hospitalization; persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions; a congenital anomaly/birth defect. Other important medical events may also, in the opinion of the Investigator, be considered SAEs. An AE was considered a TEAE if it occurred on or after the first dose, and was not present prior to the first dose, or it was present at the first dose but increased in severity during the study. Events recorded as either possibly, probably, or definitely related to treatment were categorized as related. AE severity was graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events, Version 4.03.
Time Frame: Up to 242 weeks + 30 days. SAEs were recorded beginning at the time the subject signed the informed consent form through 30 days following the last study visit. Non-serious AEs were recorded from the time of informed consent through the last study visit.
Measure: Number; unit: participants
Arm/Group | UX003
Number analyzed (Participants) | 3
participants
  Any TEAE | 3
  Treatment-related TEAE | 2
  SAE | 2
  Grade 3 or 4 TEAE | 2
  TEAE leading to treatment discontinuation | 1
  TEAE leading to study discontinuation | 0
  Fatal TEAE | 0

5. Secondary Outcome: Acceptable Dose as Determined by Total uGAG Excretion Using a Forced Dose Titration Regimen
Description: The choice of the dose of UX003 QOW for the Long-Term Extension Phase was based on a preliminary efficacy analysis at Week 36 prior to all 3 participants completing the Forced-dose Titration Period of the First Phase of the study.
Time Frame: Week 36
Measure: Number; unit: mg/kg
Arm/Group | UX003
Number analyzed (Participants) | 3
mg/kg | 4

6. Secondary Outcome: Change From Baseline at Week 36 in Six-Minute Walk Test (6MWT)
Description: The total distance walked (meters) in a 6-minute period was measured once each test day. The test was conducted using a pre-measured walking course according to administration guidelines established by the American Thoracic Society (ATS 2002). Participants who could not walk could omit this test.
Time Frame: Baseline, Week 36
Population: Summary analyses for all 3 participants are not available due to the very small number of participants; and while data were collected for 1 participant, they are not being reported due to confidentiality issues.
Arm/Group | UX003
Number analyzed (Participants) | 0

7. Secondary Outcome: Percent of Predicted Normal Distance Walked
Description: The percent of predicted normal distance walked (based on published normative data) in the total distance walked in a six-minute period.
Time Frame: 36 Weeks
Population: as for outcome 6
Arm/Group | UX003
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline at Week 36 in the 3-Minute Stair Climb Test (3MSCT)
Description: The number of stairs climbed within a 3-minute period was assessed once each test day using available hospital stairs. Participants who could not climb stairs could omit this test.
Time Frame: Baseline, Week 36
Population: as for outcome 6
Arm/Group | UX003
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline at Week 36 in Pulmonary Function Testing (Spirometry)
Description: The following spirometry tests were administered to participants who did not require invasive ventilatory support or have a tracheostomy in accordance with American Thoracic Society/European Respiratory society (ATS/ERS) guidelines: forced vital capacity (FVC), forced expiratory volume in 1 second (FEV1), maximum voluntary ventilation in one minute (MVV1). Invasive ventilation is defined as any form of ventilatory support applied with the use of an endotracheal tube.
Time Frame: Baseline, Week 36
Population: as for outcome 6
Arm/Group | UX003
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline at Week 36 in Growth Velocity for Height and Weight
Description: Growth velocity (for males ≤18 years and females ≤15) was calculated from anthropometric measurements and compared with pretreatment growth velocity when available. Z-scores and percentiles were calculated using Centers for Disease Control (CDC) growth chart.
Time Frame: Baseline, Week 36
Population: Summary analyses for all 3 participants combined are not available. Due to the very small number of participants, formal statistical analyses were not performed; and data were presented per participant, which has the potential for participant re-identification given the rarity of disease and the very small population size.
Arm/Group | UX003
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline at Week 36 in Shoulder Range of Motion (Goniometry)
Description: The maximum passive shoulder range of motion in both flexion and extension will be measured in degrees using a goniometer.
Time Frame: Baseline, Week 36
Population: as for outcome 6
Arm/Group | UX003
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Up to 242 weeks + 30 days. SAEs were recorded beginning at the time the subject signed the informed consent form through 30 days following the last study visit. Non-serious AEs were recorded from the time of informed consent through the last study visit.
Description: TEAEs are presented. An AE was considered a TEAE if it occurred on or after the first dose, and was not present prior to the first dose, or it was present at the first dose but increased in severity during the study.
Arm/Group | UX003
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | UX003 (N=3)
Inguinal hernia repair (Surgical and medical procedures) | 1
Spinal cord compression (Nervous system disorders) | 1
Cerebral ventricle dilatation (Nervous system disorders) | 1
Oedema peripheral (General disorders) | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | UX003 (N=3)
Ligament sprain (Injury, poisoning and procedural complications) | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1
Body temperature increased (Investigations) | 1
Weight increased (Investigations) | 2
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Dizziness (Nervous system disorders) | 1
Nystagmus (Nervous system disorders) | 1
Reflexes abnormal (Nervous system disorders) | 1
Visual field defect (Nervous system disorders) | 1
Discomfort (General disorders) | 1
Gait disturbance (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Generalised Oedema (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Oral mucosal erythema (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Acute sinusitis (Infections and infestations) | 1
Dermatitis infected (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Molluscum contagiosum (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Nosocomial infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Viral rash (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
This study was terminated due to business considerations unrelated to safety or efficacy concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days